CLINICAL TRIAL: NCT03281720
Title: Selective Image Guided Resection of Pathologically Documented Axillary Lymph Node Metastases
Acronym: TAD
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: UNC Lineberger Comprehensive Cancer Center (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: LCCC1622; 16-1583 (Other: UNC Chapel Hill IRB)
Record Dates: First submitted 2017-09-11; First posted 2017-09-13 (Actual); Last update posted 2023-01-04 (Actual); Status verified 2023-01

CONDITIONS: Breast Cancer
MeSH Terms: conditions — Breast Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Targeted Axillary Dissection (Experimental): After patients have completed their neoadjuvant systemic therapy, they will have a Savi Scout® electromagnetic reflector placed into the clipped axillary lymph nodes.
  The surgeon will then use the Savi Scout detector intraoperatively to identify and remove your clipped lymph nodes prior to removing the remainder of the axillary lymph nodes in a surgery called an "axillary dissection".
  Interventions: Procedure: TAD

INTERVENTIONS:
Procedure: TAD — the same intervention as listed in the arm description

SUMMARY:
The purpose of this research study is to determine how feasible and accurate identifying and removing specific lymph nodes in the axilla (armpit) after neoadjuvant systemic therapy is when patients present with breast cancer that has spread to lymph nodes in the axilla. The specific lymph nodes removed would be determined at the time of diagnosis. If a biopsy proves that cancer has spread to a lymph node, a titanium clip will placed in it to mark it for future removal. That lymph node will be removed after systemic therapy and compared with the rest of the lymph nodes removed from that region.

ELIGIBILITY:
Inclusion Criteria:

1. Histologic diagnosis of invasive breast cancer, clinical stage T0-3 N1-3 (maximum three abnormal axillary nodes on ultrasound exam) M0.
2. Core needle biopsy (or fine needle aspiration (FNA)) of an axillary node documenting nodal disease at time of diagnosis and prior to preoperative systemic therapy or surgery. Clinical care marker clip placed in the abnormal axillary nodes identified at ultrasound at the time of core needle or FNA of an axillary node that documented nodal disease.
3. Subjects must be undergoing neoadjuvant systemic therapy (or have just completed it) prior to the surgical intervention.
4. No prior axillary lymph node surgery for pathological confirmation of axillary status.
5. No nitinol (nickel-titanium) allergy. The Savi Scout ® marker device contains nitinol.
6. Females of childbearing potential must have a negative serum pregnancy test within 14 days prior to receipt of chemotherapy. NOTE: Females are considered of child bearing potential unless they are surgically sterile (have undergone a hysterectomy, bilateral tubal ligation, or bilateral oophorectomy) or they are naturally postmenopausal for at least 12 consecutive months
7. Females of childbearing potential must be willing to abstain from heterosexual activity or to use 2 forms of effective methods of contraception from the time of informed consent until 30 days after chemotherapy discontinuation. The two contraception methods can be comprised of two barrier methods, or a barrier method plus a hormonal method or an intrauterine device that meets <1% failure rate for protection from pregnancy in the product label.
8. As determined by the enrolling physician or protocol designee, ability of the subject to understand and comply with study procedures for the entire length of the study.

Exclusion Criteria:

1. Active infection requiring systemic therapy
2. Has a known additional malignancy that is active and/or progressive requiring treatment; exceptions include basal cell or squamous cell skin cancer, in situ cervical or bladder cancer.
3. Any distant metastasis by imaging and biopsy (cM1)
4. Patients not receiving neoadjuvant systemic therapy.

Ages: 18 Years to 99 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 100 (Actual)
Dates: Start 2017-04-07 (Actual); Primary Completion 2021-03-04 (Actual); Study Completion 2021-05-24 (Actual)

PRIMARY OUTCOMES:
The false negative rate of TAD | two years
  will be defined as the percentage of patients in whom the lymph nodes identified with TAD were free of residual metastatic disease while remaining metastatic disease was demonstrated in the completion axillary lymph node dissection

SECONDARY OUTCOMES:
Nodal pathologic complete response | two years
  will be defined as no residual carcinoma in any lymph node sampled during TAD and/or ALND.
The percentage of lymph nodes removed with ALND not identified by TAD that harbor residual metastasis | two years
  will be calculated by the formula: (# pos LN/# LN sampled by ALND) x 100
The success rate of preoperative localization with the Savi Scout® | two years
  will be determined by the number of reflectors placed versus the number of reflectors detected at the time of surgery.

CONTACTS AND LOCATIONS:
Locations (1):
- UNC- Chapel Hill Lineberger Comprehensive Cancer Center, Chapel Hill, North Carolina, United States